CLINICAL TRIAL: NCT01749579
Title: Comparison of Propofol-fentanyl and Midazolam-fentanyl for Conscious Sedation in Painful Procedures
Brief Title: Comparison of Propofol-fentanyl and Midazolam-fentanyl for Conscious Sedation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 130-2640
Record Dates: First submitted 2012-12-06; First posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Emergencies
Keywords: propofol; midazolam; duration of recovery; emergency procedure
MeSH Terms: conditions — Emergencies | interventions — Propofol; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Experimental): The patients will receive propofol for sedation in addition to fentanyl
  Interventions: Drug: Propofol; Drug: Fentanyl
- Midazolam (Active Comparator): The patients will receive midazolam for sedation in addition to fentanyl
  Interventions: Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol — Propofol 1 mg/kg bolus then 500 microg/kg every 2 minutes until sedation level equivalent to Ramsey 3
  Arms: Propofol
Drug: Midazolam — Midazolam 0.03 mg/Kg stat and then the same dose repeated every 2 minutes until a sedation level of Ramsey 3 is achieved.
  Arms: Midazolam
Drug: Fentanyl — Fentanyl 2 microg/kg intravenous stat and every 2 minutes until the end of procedure

SUMMARY:
Sixty patients who refer to the emergency ward and need any painful procedure in the ward are randomized into 2 groups. One group is sedated before the procedure using propofol-fentanyl and the other with midazolam-fentanyl, with the same depth of sedation. The two groups will be compared regarding recovery time and other parameters described below.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18
* candidate for a painful procedure
* negative past history of a serious medical condition
* ASA score 0 and 1

Exclusion Criteria:

* deep sedation making the patient unable to answer the questions
* pregnancy
* allergy to drugs
* hemodynamic instability
* failure to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-01 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Recovery time | Within one hour after sedation
  Length of time before complete recovery from sedation is achieved

SECONDARY OUTCOMES:
Patients' Pain perception | Within one hour after sedation
  Pain perception as measured by verbal numeric rating scale

OTHER OUTCOMES:
Blood pressure | Within one hour after sedation
Oxygen saturation | Within one hour after sedation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jalili, MD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital, Tehran, Tehran Province, Iran